CLINICAL TRIAL: NCT05983172
Title: Multi-omics Approach of Risk Stratification for Patients With de Novo Acute Myeloid Leukemia
Status: Enrolling by invitation | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Assistant Professor and attending physician, National Taiwan University Hospital
Other Study IDs: 202306138RINB
Record Dates: First submitted 2023-07-30; First posted 2023-08-09 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; Machine learning; Artificial intelligence; Risk stratification
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators will use machine learning to identify features on bone marrow smears and select features that are related to gene mutations, gene expression, or prognosis. The investigators will then use genome-wide transcriptomic profiling to investigate gene expression that is associated with patients' outcomes. The investigators will design a next-generation sequencing panel with unique molecular index and assess its feasibility and robustness in detecting measurable residual disease and optimize the panel/platform/bioinformatic pipeline. Finally, The investigators will use machine learning to integrate bone marrow smear features, gene mutations, gene expression, and measurable residual disease to construct a comprehensive risk assessment system that is based on multi-omics data. The investigators believe that such a platform will help physicians to design the most appropriate treatment strategies for individual patients, not only advancing the concept of precision medicine but also improving patients' prognoses.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with acute myeloid leukemia at the National Taiwan University Hospital
2. Ever enrolled in 201802021RINC、202109078RINB、201709072RINC

Exclusion Criteria:

Nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with acute myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of diagnosis until the date of death from any cause, assessed up to 30 years

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Cheng-Hong Tsai, MD, MSc, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No